CLINICAL TRIAL: NCT03010150
Title: Modeling Adherence to Preventive Swallowing Exercises in Head and Neck Cancer
Brief Title: Blood Tests and Questionnaires in Studying Adherence to Preventative Swallowing Exercises in Participants With Metastatic Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-0597; NCI-2018-01260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0597 (Other: M D Anderson Cancer Center); R21DE019954 (NIH)
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma of Unknown Primary; Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Metastatic Head and Neck Carcinoma; Metastatic Malignant Neoplasm in the Uterine Cervix; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Stage I Hypopharyngeal Carcinoma AJCC v8; Stage I Nasopharyngeal Carcinoma AJCC v8; Stage II Hypopharyngeal Carcinoma AJCC v8; Stage II Laryngeal Cancer AJCC v8; Stage II Nasopharyngeal Carcinoma AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Nasopharyngeal Carcinoma AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Nasopharyngeal Carcinoma AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Neoplasms, Unknown Primary; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Laryngeal Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (blood tests, questionnaires): Participants provide blood samples prior to and at the 6-month visit after receiving radiation therapy. Participants also complete questionnaires either at home, in clinic, or via internet over 30 minutes prior to receiving radiation therapy and within 14 days of blood sample collection.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Provide blood samples
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial uses blood tests and questionnaires to study how well participants with head and neck cancer that has spread to other places in the body adhere to swallowing exercises to prevent future disease. Using blood tests to study cytokines (proteins related to the immune system) may help doctors learn if certain levels of cytokines affect whether or not side effects occur and if they put participants at risk for future disease. Questionnaires may help doctors learn about the reasons head and neck cancer participants may or may not follow the swallowing exercises that they are asked to perform after receiving radiation treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether illness perceptions significantly predict adherence to swallowing exercises at 6 months after the end of radiation.

II. To determine whether sickness behaviors (depression, fatigue, pain)'s effect on illness perceptions are mediated by pro-inflammatory cytokines.

III. To determine whether social support moderates the impact of coping on appraisal of coping.

SECONDARY OBJECTIVES:

I. As a secondary aim, to determine the feasibility and utility of cardiac impedance pre-ejection period measurement as a corollary measure for depression and distress.

II. As a secondary aim, to identify potential genetic markers for swallowing dysfunction which has developed by the 6-month follow-up.

OUTLINE:

Participants provide blood samples prior to and at the 6-month visit after receiving radiation therapy. Participants also complete questionnaires either at home, in clinic, or via internet over 30 minutes prior to receiving radiation therapy and within 14 days of blood sample collection.

After completion of study, participants are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Are dispositioned to receive radiation with curative intent for nasopharyngeal, oropharyngeal, hypopharyngeal, laryngeal, or an unknown primary cancer with cervical metastases
* Are stage II-IVb for non- human papillomavirus (HPV)- related oropharyngeal cancer
* Have HPV- related oropharynx cancer that is T1, have nodal involvement with no distant metastasis or have HPV- related oropharynx cancer that is at least T2 with no distant metastasis
* Are stage II-IVb for laryngeal cancer
* Are stage I-IVb for hypopharyngeal
* Are stage I-IVb for nasopharyngeal cancer
* Have stage I-III unknown primary cancer with cervical

Exclusion Criteria:

* Have other cancer diagnoses, except non-melanoma skin cancer
* Had treatment for previous head and neck cancer or radiation to the head and neck
* Have a history of previous head and neck surgery (excluding biopsy and/or tonsillectomy and/or tracheotomy)
* Have a current oropharyngeal dysphagia unrelated to cancer diagnosis (e.g., dysphagia due to underlying neurogenic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 471 (Estimated)
Dates: Start 2016-12-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to swallowing exercises | Up to 6 months
  The primary analytic approach is to use linear mixed models to determine whether illness perceptions significantly predict adherence 6 months. The study will estimate and test the illness perception subscale scores' relationship to adherence using a linear mixed model. In the model, the dependent variable is the patient's self-reported adherence score and independent variables include illness perception, follow-up assessment time point and other covariates such as demographic and medical variables, depression, pain, fatigue, emotional coping, objective coping, appraisal of coping, stress, and lack of social well-being.
Illness perceptions | Up to 6 months
  The study's statistical tool is mediation analysis: the independent variables are the sickness behaviors (depression, fatigue, pain); the mediators are the cytokine levels, and the outcome variable is illness perception. The study will test the mediator effects based on the product of coefficients method, rather than the classical Baron & Kenny causal steps tests, since the former approach has better statistical power. The study will conduct both single-mediator analysis for each of the mediators, and multiple-mediator analysis with all mediators in the mediating process
Effect of social support on coping | Up to 6 months
  The moderating effect of social support on coping and appraisal of coping is the statistical equivalent of testing the two-way interaction between these variables and the social support variable. Multivariate linear regression will be used, in which the dependent variable is appraisal of coping at 6 months follow-up, and independent variables include the emotion-focused coping and action-focused sub scales, social support, and their two-way interactions. In the regression, the study will control for baseline variables. In addition, we will also apply the linear mixed model to investigate the moderating effect of these variables longitudinally. The mixed model naturally accounts for the correlation of repeated measures at baseline and 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H Shinn, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shinn EH, Garden AS, Peterson SK, Leupi DJ, Chen M, Blau R, Becerra L, Rafeedi T, Ramirez J, Rodriquez D, VanFossen F, Zehner S, Mercier PP, Wang J, Hutcheson K, Hanna E, Lipomi DJ. Iterative Patient Testing of a Stimuli-Responsive Swallowing Activity Sensor to Promote Extended User Engagement During the First Year After Radiation: Multiphase Remote and In-Person Observational Cohort Study. JMIR Cancer. 2024 Feb 28;10:e47359. doi: 10.2196/47359. PMID 38416544
- See also: M D Anderson Cancer Center — http://www.mdanderson.org